CLINICAL TRIAL: NCT02101099
Title: Effect of Anesthesia on Force Application During Colonoscopy
Acronym: CFM
Status: Completed | Type: Observational
Sponsor: Artann Laboratories (Industry)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH); Capital Digestive Care, LLC (Other); University of Pennsylvania (Other); Georgetown University (Other)
Responsible Party: Sponsor
Other Study IDs: CFM-04; 5R44DK068936 (NIH)
Record Dates: First submitted 2014-03-28; First posted 2014-04-01 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2016-07

CONDITIONS: Outpatient Colonoscopy for Colorectal Cancer Screening or for Symptoms Suggestive of Colonic Diseases
Keywords: Colonoscopy; Force; Monitor; Endoscopist; Conscious; Sedation; Propofol

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Patients undergoing colonoscopy: Patients who are undergoing outpatient colonoscopy for colorectal cancer screening or for symptoms suggestive of colonic diseases.
  Interventions: Device: Colonoscopy Force Monitor

INTERVENTIONS:
Device: Colonoscopy Force Monitor — Use of Colonoscopy Force Monitoring device (CFM) to measure forces applied to the colonoscope during the procedure.
  Other Names: CFM

SUMMARY:
The aim of the study is to determine if more force is used during colonoscopy when patients receive monitored anesthesia with propofol versus conscious sedation. Force measurements will be performed using the colonoscopy force monitor (CFM). This device measures the magnitude and direction of force applied to the insertion tube of a standard colonoscope during colonoscopy.

DETAILED DESCRIPTION:
Randomized factorial design of colonoscopy with either propofol administered anesthesia or conscious sedation. Twelve experienced endoscopists from community and academic centers will perform colonoscopy using either propofol or conscious sedation on a group of 12 patients for each endoscopist for a study total of 144 patients. An equal number of male and female patients will be included in each group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age: 30-75 years
* ASA Class I or II
* All ethnic and racial groups will be included

Exclusion Criteria:

* Colonic pathology that in the opinion of the endoscopist could interfere with the colonoscopy. Examples include: colonic stricture, poor preparation, obstructing tumor.
* Specific pathology that would limit the extent of examination
* ASA class 3 or greater
* Pregnancy
* Monitored anesthesia using propofol for sedation.
* Vulnerable subjects. Students, nursing home residents, institutionalized patients, and those with psychological or physical incapacity

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult male and female patients between the ages of 30 and 75 presenting to the participating sites for screening or diagnostic colonoscopy to be performed by any of the investigators will be considered for inclusion.
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2014-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Peak push force is increased in patients receiving propofol as compared to conscious sedation. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Louis Y Korman, M.D., Principal Investigator — Capital Digestive Care, LLC
Locations (3):
- United States (3):
  - Georgetown University Medical Center, Gastroenterology, Washington D.C., District of Columbia
  - Chevy Chase Endoscopy Center, Chevy Chase, Maryland
  - Univeristy of Pennsylvania Medical Center, Philadelphia, Pennsylvania